CLINICAL TRIAL: NCT05573269
Title: The Improving Effects of Fish Oil Supplementation Combined With Pine Bark Extract on Cognition in Aged-related Cognitive Decline
Brief Title: Improving Effects of Fish Oil Combined With Pine Bark Extract on Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N202012034
Record Dates: First submitted 2022-09-25; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Fish Oils; pycnogenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOPE group (Experimental): Dietary supplement, Polyphenolic extract from pine bark (Oligopin® 100mg) and fish oil capsule contained EPA 350mg + DHA 250mg. This group will receive a nutritional supplement for a period of 6 months.
  The participants will have a capsule of polyphenolic extract and a capsule of fish oil a day.
  Interventions: Dietary Supplement: FOPE (fish oil + pine extract)
- FO group (Active Comparator): This group will have placebo capsule and fish oil capsule. Placebo capsule contained maltodextrin and magnesium stearate, while fish oil contained EPA 350mg + DHA 250mg. The participants will receive the supplements for a period of 6 months and have a capsule of placebo and a capsule of fish oil a day.
  Interventions: Other: FO (fish oil +placebo)

INTERVENTIONS:
Dietary Supplement: FOPE (fish oil + pine extract) — During the experiment period the participants will receive a capsule of pine bark extract (Oligopin® 100mg) and a capsule of fish oil (EPA 350mg + DHA 250mg) a day. Blood collecting (biomedical parameters and antioxidative status) and cognitive function evaluation will be examined at the 0, 12, 24th week. Body composition, 24-hour dietary recall and blood pressure measurement will be measured at 0, 4, 8, 12, 16, 20, 24th week.
  Arms: FOPE group
Other: FO (fish oil +placebo) — During the experiment period the participants will receive a capsule of placebo (maltodextrin + magnesium stearate) and a capsule of fish oil (EPA 350mg + DHA 250mg) a day. Blood collecting (biomedical parameters and antioxidative status) and cognitive function evaluation will be examined at the 0, 12, 24th week. Body composition, 24-hour dietary recall and blood pressure measurement will be measured at 0, 4, 8, 12, 16, 20, 24th week.
  Arms: FO group

SUMMARY:
The purpose of this study is to evaluate the improving effects of ω-3 fatty acid from fish oil combined with polyphenolic extract from pine bark (PE) on cognitive functions and biological parameters in healthy people aged 55 to 75.

DETAILED DESCRIPTION:
Sixty participants who meet the inclusion criteria will be randomly divided into two groups. Participants in FO group will be provided one capsule of fish oil (350mg EPA + 250mg DHA) per day for 6 months. Moreover, participants in FOPE group will be provided one capsule of fish oil (350mg EPA + 250mg DHA) combined with PE (100mg Oligopin) per day for 6 months. A cognitive function evaluation, blood biological analysis and antioxidative status will be carried out at the baseline, 3 th month and the end of the supplementation period. On the other hand, blood fatty acid composition will be measured at the baseline and the end of the supplementation period. All participants will come to laboratory and receive the supplements every month. At the same time, they will accept the measurement of body weight and blood pressure, also be interviewed with 24 hours dietary recall questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* I. 55~75 years old
* II. No severe diseases, such as hyperlipidemia, diabetes, heart diseases, cancer etc.
* III. Mini-mental state examination (MMSE) score is more than 26
* IV. Clinical dementia rating scale (CDRS) score is less than 0.5

Exclusion Criteria:

* liver disease, kidney disease, hypertension, hyperlipidemia, anemia, cancer

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  The most commonly used cognitive function assessment tool in clinical.
Clinical Dementia Rating Scale (CDRS) | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  CDR is a rating scale for staging patients diagnosed with dementia. no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2), and severe cognitive impairment (CDR = 3)
Cognitive Ability Screening Instrument (CASI) | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  CASI is a cognitive test screening for dementia. For monitoring the disease progression and providing profiles of cognitive impairment by examining abilities on attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, list-generating fluency and abstraction.

SECONDARY OUTCOMES:
Liver function -AST | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum AST is in units per liter.
Liver function -ALT | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum ALT is in units per liter.
Kidney function -BUN | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum BUN is in milligram per deciliter
Kidney function -Creatine | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum creatine is in milligram per deciliter
Kidney function -uric acid | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum uric acid is in milligram per deciliter
Lipid profile | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum HDL-Cho, LDL-Cho, triglyceride and total cholesterol are in milligram per deciliter
An outcome related with hematology- white blood cell related measurements | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum WBC in 1000/uL; neutrophils, lymphocytes, monocytes, eosinophils and basophils are in percentage.
An outcome related with hematology- red blood cell related measurements | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  RBC in 1000000/uL
An outcome related with hematology- platelet | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Platelet in 1000/uL
Nutritional status | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Serum albumin is in gram per deciliter
Antioxidative status -TBARS | Change from Baseline at the 12th and 24th week
  Thiobarbituric acid-reactive substance
Antioxidative status -GSH/GSSG | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  glutathione/oxidized glutathione ratio
Antioxidative status-Oxidized LDL | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Oxidized LDL
Antioxidative status-SOD | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Superoxide dismutase
Lipid composition on red blood cell membrane | Change from Baseline and the 12th and 24th week, the experiment will least for 6 months
  Lipid composition on the cell membrane of red blood cell. It will be analyzed by GC/MS system and based on the protocol of Wang et al. The composition of C16:0, C18:0, C18:1, C18:2, C18:3, C20:4, C20:5, C22:5, C22:6, saturated fatty acids, polyunsaturated fatty acids, monounsaturated fatty acids, total n-3 fatty acids, total n-6 fatty acids and the ratio of n-3 and n-6 will be measured.
  C16:0, C18:0, C18:1, C18:2, C18:3, C20:4, C20:5, C22:5, C22:6, saturated fatty acids, polyunsaturated fatty acids, monounsaturated fatty acids, total n-3 fatty acids, total n-6 fatty acids are in percentage.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Taiwan Adventist Hospital, Taipei